CLINICAL TRIAL: NCT01783288
Title: Aldosterone and Sodium Regulation in Postural Tachycardia Syndrome - Screening Protocol
Brief Title: Aldosterone & Sodium Regulation in Postural Tachycardia Syndrome - Screening
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Alfredo Gamboa, Research Associate Professor of Medicine, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: IRB 121817; R01HL102387 (NIH)
Record Dates: First submitted 2013-01-25; First posted 2013-02-04 (Estimated); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Postural Tachycardia Syndrome
Keywords: Postural tachycardia syndrome; orthostatic intolerance; orthostatic tachycardia; POTS
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome; Orthostatic Intolerance | interventions — Supine Position; Heart Rate; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All participants (Other): All participants will be administered all procedures as described previously.
  Interventions:
  Autonomic Function Testing, Posture Study ,Measurement of Total Blood Volume ,Exercise Capacity Test
  Interventions: Other: Autonomic Function Testing; Other: Posture Study; Procedure: Measurement of Total Blood Volume; Other: Exercise Capacity Test

INTERVENTIONS:
Other: Autonomic Function Testing — heart rate and blood pressure will be continuously monitored while participants undergo a variety of breathing techniques (deep breathing, rapid breathing, blowing against resistance) and during sustained handgrip and cold pressor (hand in ice water). All tests are meant to stimulate the autonomic nervous system to produce changes in blood pressure and heart rate of short duration that reflect how well the autonomic nervous system is functioning.
  Also during autonomic function testing, cardiac output will be measured to analyze the shift of fluids in the body (body impedance) and / or by analyzing the air that is breathed.
Other: Posture Study — Blood pressure, heart rate and blood samples (for catecholamines and hormones) will be measured & collected in the supine (lying) and upright position for each participant.
  Other Names: Supine & standing blood pressure, heart rate & blood draws.
Procedure: Measurement of Total Blood Volume — Total blood volume is measured by using iodinated I-131 tagged human serum albumin.
  Other Names: blood sample at baseline and at 12 minutes; I-131 is administered.
Other: Exercise Capacity Test — Participants will ride on a stationary recumbent bicycle and the resistance will be gradually increased while expired air is measured.
  Other Names: Masimal Oxygen Consumption Test

SUMMARY:
The purpose of the study is to determine whether patients meet criteria for Postural Tachycardia Syndrome (or not) and have reduced blood volume (or not). Both of these are important screening elements to Aim 3 of a National Institutes of Health Grant. The purposes of Aim 3 are to determine 1. whether a high dietary sodium level appropriately expands plasma volume in Postural Orthostatic Tachycardia, 2. whether plasma renin activity and aldosterone are modified appropriately by changes in dietary sodium in Postural Tachycardia Syndrome and 3. whether patients with Postural Tachycardia Syndrome have improvements in their orthostatic tachycardia and symptoms as a result of a high dietary sodium level.

DETAILED DESCRIPTION:
The protocol consists of a screening visit and evaluation of their autonomic nervous system status. The following activities are part of this study. Subjects may stay for 2 nights and 3 study days.

Day 0 Participants will be admitted to the Clinical Research Center, their medical history, physical exam, routine lab work (hemoglobin/hematocrit & CMP) and a serum pregnancy test will be done during that first day. They will also be asked to fill out a health questionnaire. Later that day they will be evaluated to determine the extent of fatigue, depression and anxiety ratings, autonomic symptoms and quality of life, with the use of questionnaires.

Subjects may be asked to stop taking some medications for up to 7 days; it will be decided on an individual basis and after considering each medication and its effect to the autonomic nervous system. If subjects are asked to discontinue the medication, they will ask them to keep a diary of symptoms and to contact the PI or staff by phone if any new symptom appears. If necessary, medications will be restarted.

Testing day 1:

In the morning during the posture test, 5 teaspoons of blood will be drawn while subject is lying down, and after sitting and or standing for 30 minutes to measure substances produced by the body in response to inflammation and oxidative stress and to determine hormones that regulate the blood pressure. Blood pressure and heart rate will be measured in these different positions. A total of 10 tablespoons will be drawn.

In the afternoon, more tests will be performed designed to determine how well the autonomic nervous system is working in regulating blood pressure and heart rate. Autonomic function test will be performed to see how the involuntary nervous system is working. For these tests, heart rate will be recorded using a continuous electrocardiographic trace, blood pressure using a cuff around one arm and/or finger and heart's pumping capacity (cardiac output) will be measured by analyzing the shift of fluids in the body (body impedance) and/or by analyzing the air that is breathe.

Participants will be tilted up on a tilt table for 10 minutes while recording their heart rate and blood pressure. The autonomic function tests include asking the participants to breathe deeply for two minutes and breathing rapidly for 30 seconds, maintaining a handgrip for 3 minutes, blowing against pressure for 15 seconds and placing one hand in ice water for 1 minute. All these tests are meant to stimulate the autonomic nervous system to produce changes in blood pressure and heart rate of short duration that reflect how well the involuntary nervous system is working.

Testing day 2:

In the morning, total blood volume will be measured by using iodinated I-131 tagged human serum albumin, a material with a very small amount of radioactive substance. The test involves drawing a blood sample before the I-131 is given, then giving the I-131 through a catheter in one vein, waiting 12 minutes before the second blood sample is drawn to check its concentration. Blood samples will also be drawn while subjects are lying down to measure for hormones, which control blood pressure and heart rate. Blood will drawn at several points during the study. The total amount of blood drawn during this study is approximately 3 teaspoons.

In the afternoon, exercise capacity test with estimation of maximal oxygen consumption (VO2 max) will be done. This test will be conducted on a stationary bicycle and the resistance will be gradually increased while the expired air is measured during exhaustive physical work. The test will last approximately 30 minutes. A mouthpiece with a one way re-breathing valve attached to a breathing tube will be used to collect air samples during the exercise test. Essentially, subjects will breathe room air through a mouthpiece, and then expire the air into a tube that connects to a machine (metabolic cart). This machine analyzes carbon dioxide and oxygen content, which allows us to calculate the amount of oxygen they are using under resting and exercise conditions.

The workload will be gradually increased on the bike by increasing the resistance. As the workload increases, oxygen consumption also increases. Throughout the test period exhaled air will be collected. When subjects can no longer continue, the test will be stopped. Blood pressure will be measured at the end of each resistance-stage. Heart rate data will be recorded continuously.

Before and after completing the exercise test, subjects will be required to complete a "warm-up" and "cool-down" session including stretching exercises.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-50 years old
* Patients with suspected POTS and healthy volunteers
* Sedentary healthy subjects of similar age and gender than patients will also be recruited.
* Only female participants are eligible.
* Able and willing to provide informed consent

Exclusion Criteria:

* Smokers
* Overt cause for postural tachycardia, i.e., acute dehydration
* Significant cardiovascular, pulmonary, hepatic, or hematological disease by history or prior testing
* Highly trained athletes
* Subjects with somatization or severe anxiety symptoms will be excluded
* Pregnant (positive pregnancy test) or breastfeeding
* Hypertension defined as supine resting BP>145/95 mmHg off medications or needing antihypertensive medication
* Other factors which in the investigator's opinion would prevent the participant from completing the protocol, including poor compliance during previous studies or an unpredictable schedule
* Unable to give informed consent

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Estimated)
Dates: Start 2013-02 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
blood volume deviation (%) from individual predicted volumes | 2 days
  Compare blood volume deviations using the 131-I-Albumin method. Deviations will be reported as a percentage deviation from an individual's predicted value. These values will be compared between POTS patients and healthy control groups.

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo J Gamboa, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States